CLINICAL TRIAL: NCT05697926
Title: Preclinical Research for Personalized TCR-T Therapy for Head and Neck Cancer
Status: Recruiting | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022105
Record Dates: First submitted 2023-01-01; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Head and Neck Cancer
Keywords: TCR-T therapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experiment: The excess tumor tissue from patients following surgical resection will be collected for further analysis.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a preclinical study. No intervention will be performed.

SUMMARY:
This study will obtain tumor samples from patients with head and neck cancers and aims to develop personalized TCR-T therapy for head and neck cancer by determining the reactive TCR clone sequences in head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Gender is not limited, age 18-75 years old;
2. Estimated survival is greater than 3 months;
3. Newly diagnosed patients with head and neck cancer without any treatment, or patients with refractory recurrent advanced head and neck cancer for which there is no available effective treatment;
4. Patients with head and neck cancer whose tumor tissue can be surgically harvested;
5. Volunteer to join the study and sign the informed consent.

Exclusion Criteria:

1. Infected or had been infected with COVID-19;
2. Active hepatitis B or C virus, HIV infection, or other uncured active infected persons;
3. Patients with head and neck cancer who had received the following treatments:

   The patient had a history of using PD-1 and other immune checkpoint inhibitors 8 weeks before surgery; History of chemotherapy drug use 8 weeks before surgery; A history of hormone drug use within 4 weeks before surgery;
4. Other situations that are not appropriate to be included in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients with head and neck cancer without any treatment and willing to take part in this preclinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical prognosis | 5 year postsurgery
  Observation of the clinical prognosis including overall survival, progression-free survival, event-free survival, and recurrence-free survival.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China